CLINICAL TRIAL: NCT01393093
Title: Clinical Trial of Transcatheter Arterial Chemoembolization With KMG Microsphere Treating Advance-stage Hepatocellular Carinomas
Brief Title: Transcatheter Arterial Chemoembolization With KMG Microsphere Treating Advance-stage Hepatocellular Carinomas
Acronym: TACE-KMG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TMU-CIH-IR-002
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2010-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TACE -oil (Active Comparator): embolization agent:Iodinated Oil or /and gelatin sponge Iodinated Oil （5-30ml）with Epirubicin （30-40mg/m2） or and gelatin sponge
  Interventions: Procedure: Therapeutic Chemoembolization
- TACE-KMG ( routine dose Chemo) (Experimental): embolization agent:KMG microsphere( 150-450µm,0.2-2g) with routine dose Epirubicin （30-40mg/m2）
  Interventions: Procedure: Therapeutic Chemoembolization
- TACE-KMG( low dose Chemo ) (Experimental): embolization agent:KMG microsphere( 150-450µm,0.2-2g) with low dose Epirubicin （5-10mg/m2）
  Interventions: Procedure: Therapeutic Chemoembolization
- TACE-KMG(withou chemo) (Experimental): embolization agent:KMG microsphere( 150-450µm,0.2-2g)
  Interventions: Procedure: Therapeutic Chemoembolization

INTERVENTIONS:
Procedure: Therapeutic Chemoembolization — Transcatheter Arterial Chemoembolization
  Other Names: Transcatheter Arterial Chemoembolization，TACE

SUMMARY:
The purpose of the study is to evaluate the effects of Transcatheter Arterial Chemoembolization (TACE) with KMG microsphere in treating advance-stage Hepatocellular Carinoma(HCC).

DETAILED DESCRIPTION:
This is a prospective, multicentre, random, controlled clinical trial of Transcatheter Arterial Chemoembolization (TACE)with KMG Microsphere Treating Advance-stage Hepatocellular Carinomas.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular Carinomas with diagnosis of pathology or cytology or consistent with China 2001 guideline of Clinical Diagnosis Hepatocellular Carinomas
2. clinical stage（The Barcelona Liver Clinic staging system,BCLC B and C)，or can not receive surgical intervention
3. liver function:Child-Pugh A、B
4. PST 0-1（Eastern Cooperative Oncology Group Performance Score ,ECOG）
5. Lifespan≥6 months
6. First time to receive treatment
7. Can accept the follow up
8. informed consent was gotten
9. the number of lesion ≤ 5

Exclusion Criteria:

1. pregnant or lactation woman
2. emotional disturbance
3. serious heart ,lung disfunction or serious diabetes mellitus
4. serious reactiveness infections;（exp:type B or C hepatitis）
5. liver function :Child-Pugh Score C
6. thrombocyte<6×109/L
7. diffuse HCC
8. widespread metastasis
9. serious atherosclerosis
10. acquired immunodeficiency syndrome;AIDS
11. thrombosis or thrombosis event in 6 months
12. renal inadequacy who need hemodialysis or peritoneal dialysis
13. with other tumors except basal cell carcinoma and carcinoma in situ of cervix
14. serious alimentary tract hemorrhage in 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2840 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-11 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 3 years
  Time to progression

SECONDARY OUTCOMES:
total survival | 3 year
  total survival
remission rate | 3 years
  remiision rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Guo, MD, Study Chair — Tianjin Medical University Cancer Hospital
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- See also: Related Info — http://www.tjmuch.com/